CLINICAL TRIAL: NCT04517955
Title: TAVI in Intermediate Risk Septuagenarians With Risk Factors Not Captured by the Traditional Surgical Risk Scores
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor of Cardiology, University of Athens
Other Study IDs: 088891/2019
Record Dates: First submitted 2020-08-10; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: aortic stenosis; TAVI; Evolut R; Evolut Pro
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Transcatheter Aortic Valve Implantation with Evolut R or Evolut Pro
  Other Names: Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
Single arm, observational trial of Transcatheter Aortic Valve Implantation (TAVI) with the Medtronic Evolut R and Evolut Pro The primary objective of this trial is to evaluate device success of TAVI with the Evolut R and Evolut Pro systems in septuagenarians with risk factors for adverse surgical outcomes not captured by the traditional risk scores and therefore of intermediate surgical risk.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and efficacy of transcatheter aortic valve implantation (TAVI) in septuagenarians with severe, symptomatic Aortic Stenosis (AS) and risk factors for adverse surgical outcomes not captured by the traditional risk scores and therefore of intermediate surgical risk.

The primary objective of this trial is to evaluate device success of TAVI with the Evolut R and Evolut Pro systems in septuagenarians with risk factors for adverse surgical outcomes not captured by the traditional risk scores and therefore of intermediate surgical risk.

The secondary objective is to assess early safety (at 30 days) and clinical efficacy (after 30 days) of the TAVI procedure.

Exploratory objective: comparative health economics in septuagenarians with symptomatic severe aortic stenosis and intermediate surgical risk treated with Transcatheter Aortic Valve Implantation (TAVI) vs Surgical Aortic Valve Replacement (SAVR) (matched historic cohort)

ELIGIBILITY:
Inclusion Criteria:

1. Age 75-79
2. Subject must have Society of Thoracic Surgeons (STS) score >=4% and <=8%
3. Subject must have at least one from the risk factors presented below:

   i. Severely atherosclerotic or porcelain aorta ii. Internal Mammary Artery (IMA) or other conduit(s) crossing midline and/or adherent to posterior table of sternum iii. Pre-existing mechanical valve in any other position iv. Severe right ventricular dysfunction v. Hostile chest (abnormal chest wall anatomy due to severe kyphoscoliosis or other skeletal abnormalities, evidence of severe radiation damage, history of multiple recurrent pleural effusions causing internal adhesions) vi. Severe liver disease/cirrhosis vii. Frailty viii. Malignancy with life expectancy that exceeds 24 months ix. Renal replacement therapy with creatinine levels >200mmol/L or 2.26 mg/dl
4. Heart team consisting of at least one interventional cardiologist and one cardiac surgeon agree on indication and treatment proposal, based on their clinical judgment (including anatomy assessment, risk factors, etc)
5. Critical aortic valve area defined as an initial aortic valve area of <=1cm2 or aortic valve index <0.6cm2/m2
6. In presence of normal left ventricular function:

   1. Mean gradient >40mmHg OR Vmax>4m/sec OR
   2. In presence of low flow, low gradient severe AS, a dobutamine stress echo must be conducted that demonstrates presence of contractile reserve defined as follows >=20% increase in stroke volume and mean gradient >40mmHg
7. Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater
8. The subject is suitable for direct TAVI not preceded by balloon valvuloplasty according to the judgment of the treating physicians
9. The subject and the treating physician agree that the subject will return for all required post procedure follow-up visits.

Exclusion Criteria:

1. Hypersensitivity or contraindication to aspirin, heparin, clopidogrel, coumadin, nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated;
2. Blood dyscrasias as defined: leukopenia (WBC<1000/mm3), thrombocytopenia (platelet count <50.000cells/mm3), history of bleeding diathesis or coagulopathy;
3. Ongoing sepsis, including active endocarditis
4. Any condition considered a contraindication to extracorporeal assistance;
5. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within six weeks prior treatment
6. Cardiogenic shock manifested by low cardiac output, vasopressor dependence or mechanical hemodynamic support;
7. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
8. Active gastrointestinal (GI) bleeding within the past 3 months
9. Subject refuses a blood transfusion;
10. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits);
11. Multivessel coronary artery disease with a Syntax score >22
12. Estimated life expectancy of less than 24 months due to associated non-cardiac comorbid conditions
13. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consentor adherence to the protocol required follow-up exams;
14. Currently participating in an investigational drug or another device trial (excluding registries)
15. Evidence of an acute myocardial infarction <=30 days before the index procedure
16. Need for emergency surgery for any reason
17. Uncontrolled atrial fibrillation

    Anatomical Exclusion Criteria:
18. Native aortic annulus size <18mm or >30mm per the baseline diagnostic imaging;
19. Mixed aortic valve disease [aortic stenosis and aortic regurgitation with predominant aortic regurgitation (3-4+]
20. Severe mitral or severe tricuspid regurgitation
21. Severe mitral stenosis;
22. Hypertrophic obstructive cardiomyopathy
23. Echocardiographic or Multislice Computed Tomography (MSCT) evidence of intracardiac mass, thrombus or vegetation
24. Anatomy of the aortic root and ascending aorta not suitable for TAVI with Evolut R or Evolut Pro system (aortic root angulation >70 degrees for femoral and left subclavian access or >30 degrees for right subclavian access)
25. Congenital bicuspid or unicuspid valve verified by echocardiography Vascular Exclusion Criteria
26. Transarterial access not able to accommodate an 16 French sheath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 75-79 years old who have symptomatic severe aortic stenosis at intermediate surgical risk defined by a Society of Thoracic Surgeons (STS) mortality risk of >=4% and <=8%, will be presented to the Heart Team for inclusion in the trial.
  Patients will have risk factors not captured by traditional risk scores
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Device success (VARC-2 criteria) | 30 days
  1. Absence of procedural mortality
  2. Correct positioning of the prosthetic heart valve into the proper anatomical location
  3. Intended performance of the prosthetic heart valve (mean aortic valve gradient<20mmHg or peak velocity < 3m/s, and no moderate or severe prosthetic valve regurgitation) as assessed with 24h post implantation and pre-discharge echocardiogram

SECONDARY OUTCOMES:
Rate of All-cause mortality | 30 days
  Early Safety
Rate of All stroke (disabling and non-disabling) | 30 days
  Early Safety
Rate of Life-threatening bleeding | 30 days
  Early Safety
Rate of Acute Kidney Injury-Stage 2 or 3 (including renal replacement therapy) | 30 days
  Early Safety
Rate of Coronary artery obstruction requiring intervention | 30 days
  Early Safety
Rate of Major vascular complication | 30 days
  Early Safety
Rate of Valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVR) | 30 days
  Early Safety
Rate of New pacemaker implantation | 30 days
  Early Safety
Rate of All-cause mortality | after 30 days and up to 2 years
  Clinical Efficacy
Rate of All stroke (disabling and non-disabling) | after 30 days and up to 2 years
  Clinical Efficacy
Rate of Hospitalizations for valve-related symptoms or worsening congestive heart failure NYHA class III or IV | after 30 days and up to 2 years
  Clinical Efficacy
Rate of Valve related dysfunction | after 30 days and up to 2 years
  Mean aortic valve gradient >=20mmHg, Effective orifice area (EOA)<=0.9-1.1cm2, and/or Dimensionless Valve Index (DVI)<0.35 m/s and/or moderate or severe prosthetic valve regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, Prof, Principal Investigator — First Department of Cardiology, University of Athens
Locations (5):
- Greece (5):
  - Cardiology Department, Hippokration Hospital, Athens
  - First Department of Cardiology, National & Kapodistrian University of Athens, Athens
  - Onassis Cardiac Surgery Center, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina

IPD SHARING:
Plan to Share IPD: Undecided